CLINICAL TRIAL: NCT05930015
Title: Effects of Music Combined With Sports Games on Alleviating Psychological Stress, Anxiety and Mental Energy Among Adolescents During COVID-19 Pandemic in Lanzhou Gansu Province China (phase2) Research Object 1 To Develop a Music and Sports Games Program for the Secondary School-aged Adolescents. 2 To Examine the Time Effects (Within Groups), Groups Effects (Between Groups) and Interaction Effects (Within-between Groups) of Music and Sports Games on Stress, Anxiety, Mental Energy, Mental Toughness, Self-efficacy and Emotions Among Secondary Schoolaged Adolescents in GanSu Province China.
Brief Title: Effects of Music Combined With Sports Games on Alleviating Psychological Stress, Anxiety and Mental Energy Among Adolescents During COVID-19 Pandemic in Lanzhou Gansu Province China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wu Jiarun (Other)
Responsible Party: Sponsor-Investigator, Wu Jiarun, student, Universiti Sains Malaysia
Organization: Universiti Sains Malaysia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WJiarun
Record Dates: First submitted 2023-07-01; First posted 2023-07-05 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-07

CONDITIONS: Stress; Anxiety and Fear
Keywords: Stress, anxiety and fear of COVID-19
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The 200 people tested were randomly divided into 4 groups of 50 each during the intervention phase, with three groups carrying out a intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Music intervention only (Experimental): Music only (the fast tempo of 120-130 bpm music will be selected) The effect was achieved by playing music selected by the researchers during originally physical education classes in school.
  Interventions: Behavioral: Music intervention only
- Sports games intervention only (Experimental): Sports games intervention only The effect was achieved by replacing the school's originally physical education classes with sports games of the researchers' choice.
  Interventions: Behavioral: Sports games intervention only
- Music and sports games intervention (Experimental): Music and sports games intervention, the effect was achieved by replacing the school's physical education classes with sports games of the researchers' choice, and then by playing music of the researchers' choice during class.
  Interventions: Behavioral: Music and sports games intervention

INTERVENTIONS:
Behavioral: Music intervention only — Music only (120-130 bpm) The effect was achieved by playing music selected by the researchers during originally physical education classes in school; twice a week for eight weeks
  Arms: Music intervention only
Behavioral: Sports games intervention only — Sports games intervention only The effect was achieved by replacing the school's originally physical education classes with sports games of the researchers' choice; twice a week for eight weeks
  Arms: Sports games intervention only
Behavioral: Music and sports games intervention — Music and sports games intervention, the effect was achieved by replacing the school's physical education classes with sports games of the researchers' choice, and then by playing music of the researchers' choice during class; twice a week for eight weeks
  Arms: Music and sports games intervention

SUMMARY:
The objective of this observational study was to assess whether music and sports play interventions were effective in reducing stress, anxiety and fear of COVID-19 among secondary school students in Gansu Province; The effects of music, sports games, and music combined with sports games were compared.

ELIGIBILITY:
Inclusion Criteria:

* 1. Secondary schools' students (both maile and female) in Lanzhou city, years (14-17 years old).
* 2. Able to read and understand the Chinese version questionnaires.
* 3. Understand the information explained by the researcher and agree to be included in the study.
* 4. They are in good health, measured by PAR-Q
* 5. Participants who written consent to participate in the study.

Exclusion Criteria:

* Participants with disabilities that prevent them from physically active. Also, those who withdraw in the middle or at the end of the intervention before answering the questionnaire of post-trial.

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2022-12-10 (Actual); Study Completion 2022-12-10 (Actual)

PRIMARY OUTCOMES:
Change from the Stress and anxiety to viral epidemics-6 (SAVE-6) at week 8 | week 8
  Save-6 is a questionnaire developed by South Korean scholars Chung et al. (2021) in 2021 to measure the stress and anxiety responses of ordinary residents to COVID-19. The questionnaire contains six questions, including six major symptoms of stress and anxiety in the general public in response to COVID-19. The save-6 scale obtained good internal consistency after use in Korea (Cronbach's Alpha = 0.815). The Save-6 scale was found to be a reliable, valid and useful simple measurement that could be applied to the general population.
Change from the Fear of COVID-19 scale (FCV-19) at week 8 | week 8
  The Fear of Coronavirus Scale is a questionnaire designed to measure the Fear, concern and anxiety of the general public regarding COVID-19. It was developed by Ahorsu et al. (2020) research and development. The questionnaire includes seven items of public fear of COVID-19 (item-total correlation (0.47 to 0.56)). More specifically, Reliability values such as internal consistency (α =.82) and test -- retest reliability (ICC =.72) were acceptable. The Fear of COVID-19 Scale, a seven-item scale, has robust psychometric properties. It is reliable and valid in assessing fear of COVID-19 among the general population and will also be useful in allaying COVID-19 fears among individuals.

SECONDARY OUTCOMES:
Change from the Athletic Mental Energy Scale (AMES) at week 8 | week 8
  Athletic Mental Energy Scale (AMES) is a questionnaire developed by Lu et al. (2018) which is specially used to measure Mental Energy. The questionnaire consists of 18 related questions. The test subjects need to choose the most consistent level from the six feelings (completely so - completely not) according to their feelings, and each feeling has corresponding score (6-1). The final score can represent the mental energy of the subject. The questionnaire obtained high reliability (Cronbach's α = 0.95) after being used in Taiwan and Malaysia, and proved to be an effective mental energy measurement tool.
Change from the Mental Toughness Questionnaire (MTQ) at week 8 | week 8
  Clough et al. (2002) developed a measure of mental toughness known as the Mental Toughness Questionnaire-48 (MTQ-48). The questionnaire contains 48 questions about mental toughness. Participants were asked to choose the most consistent of five feelings (strongly disagree - strongly agree) based on how they felt, with each feeling given a score (1-5). The final score represents the participants' mental toughness. The questionnaire has been widely used to measure mental toughness and is an effective measurement tool.
Change from the Portuguese Physical Literacy Assessment Questionnaire (PPLA-Q) at week 8 | week 8
  Portuguese Physical Literacy Assessment Questionnaire (PPLA-Q) is a survey published by Mota et al. (2021). The developed questionnaire is designed to measure the physical literacy of high school students. The questionnaire contains three modules of cognitive, psychology and social. In this study, we choose the module of psychological (46 likert-type items). Participants were asked to choose the most consistent of five feelings (not at all - totally) based on how they felt, with each feeling given a score (0-4). The final score represents the participants' Physical literacy. The questionnaire has been used to measure middle school students in Portugal and is an effective measurement tool.
Change from the Achievement Emotions Adjective List (AEAL) at week 8 | week 8
  The Achievement Emotions Adjective List (AEAL) is a brief self-report multi-item questionnaire deputed to assess ten achievement emotions, namely enjoyment, pride, hope, relief, relaxation, anxiety, anger, shame, hopelessness, and boredom. The AEAL is a questionnaire developed by Raccanello et al. (2021) and it scale achieved good internal consistency after use in Switzerland's middle school students (Cronbach's Alpha = 0.78). AEAL is considered to be a simple, non-invasive and effective tool for assessing the emotions of middle school students.
Saliva cortisol levels | week 8
  Saliva cortisol levels should be measured according to the tools and methods required by local medical institutions. Saliva of some subjects should be collected and handed over to local medical institutions for relevant measurement.
Heart rate variability (HRV) | week 8
  HRV data were collected using a heart rate variability (HRV) analyser.
Blood oxygen saturation (SaO2) | week 8
  Blood oxygen saturation (SaO2) data were collected using an oxygen saturation tester.

CONTACTS AND LOCATIONS:
Locations (1):
- Universiti Sains Malaysia, Kota Bharu, Kelantan, Malaysia